CLINICAL TRIAL: NCT03698604
Title: Total Laparoscopic Hysterectomy Versus Total Abdominal Hysterectomy in Women With Endometrial Neoplasia; Randomized Controlled Clinical Trial
Brief Title: Total Laparoscopic Hysterectomy Versus Total Abdominal Hysterectomy in Women With Endometrial Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Rania Gamal Anwar Elskaan, Assistant Lecturer, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLH-TAH-EN
Record Dates: First submitted 2018-09-26; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Hysterectomy; Laparoscopy
MeSH Terms: interventions — Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Laparoscopic Hysterectomy (Active Comparator): The group that will undergo total laparoscopy hysterectomy with bilateral salpingoophrectomy.
  Interventions: Procedure: Hysterectomy
- Total Abdominal hysterectomy (Active Comparator): The group that will undergo total abdominal hysterectomy with bilateral salpingoophrectomy.
  Interventions: Procedure: Hysterectomy

INTERVENTIONS:
Procedure: Hysterectomy — Total Laparoscopic Hysterectomy Total Abdominal hysterectomy

SUMMARY:
The aim of this study is to compare operative time between total laparoscopy hysterectomy with bilateral salpingoophrectomy (TLH+BSO) versus total abdominal hysterectomy and bilateral salpingooophorectomy (TAH+BSO) in women with uterine neoplasia.

DETAILED DESCRIPTION:
Research Questions:

Is total laparoscopic hysterectomy associated with similar operative operative time as total abdominal hysterectomy and bilateral salpingoophrectomy in women with uterine neoplasia?

Research Hypothesis:

In women with uterine neoplasia TLH with BSO may be similar to TAH with BSO as regard operative time.

ELIGIBILITY:
Inclusion Criteria:

The presence of perimenopausal bleeding

* Early stage endometrial carcinoma.
* Endometrial hyperplasia with/without atypia.

Exclusion Criteria:

* Obese patients i.e., BMI< 29 k.g/m2.
* Patients unfit for laparoscopy as patients with cardio-pulmonary compromise.
* Presence of adnexal mass.
* End stage endometrial carcinoma stage 3 & 4.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Operative time | From skin incision till closure of the vault "up to 4 hours".
  Operative time measured in minutes using stopwatch excluding time of concomitant surgical procedures.

SECONDARY OUTCOMES:
Blood loss | From skin incision start until skin suturing is finished "up to 4 hours".
  Intra operative blood loss will be estimated via:
  1. Amount of blood in the suction bottle.
  2. Estimation will be based on number of soaked gauzes and towels (soaked gauze = 20 ml blood; soaked towel = 150 ml; semi soaked towel = 75 ml).
Blood transfusion | From admission to the hospital until the home discharge "up to 1 week".
  The need to blood transfusion to the patient.
Postoperative pain | 8 hours after the end of operation.
  Assessment of pain intensity using Visual Analog Scale (VAS) which is one-dimensional measure of pain intensity.
  It is a continuous scale comprised of a horizontal line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. The scale is anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100).
Hospital stay | From admission to the hospital until the home discharge "up to 1 week".
  Hospital stay duration in days.
Incidence of operative complications | During operation.
  The need for laparotomy, and bowel or bladder or ureteric injury.
Incidence of postoperative complications | Up to 1 week postoperative.
  Morbidities e.g.:
  * Vaginal vault hematoma or pelvic hematoma or abscess.
  * Surgical site infection.
  * Urinary tract infection.
  * Need for post-operative blood transfusion.
  * Postoperative bowel or urinary tract complications.

CONTACTS AND LOCATIONS:
Overall Officials: Walid E Mohammed, MD, Study Director — Ain Shams Maternity Hospital; Mortada E Ahmed, MD, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt